CLINICAL TRIAL: NCT03368781
Title: Utilizing Novel Dipole Density Capabilities to Objectively Visualize the Etiology of Recurrent Atrial Fibrillation Following a Failed AF Ablation (RECOVER AF)
Brief Title: AcQMap Objectively Visualize the Etiology of Recurrent AF Following a Failed AF Ablation
Acronym: RECOVER AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP-AF-004; CLP-AF-005 (Other: Acutus Medical); CLP-AF-004-NL (Other: Acutus Medical, Inc.); NCT03467126 (obsolete NCT alias)
Record Dates: First submitted 2017-12-01; First posted 2017-12-11 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: None randomized, single-arm, open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AcQMap Imaging and Mapping (Experimental): Use of the AcQMap Imaging and Mapping System as a diagnostic modality in an ablation retreatment procedure for recurrent atrial fibrillation following a failed AF ablation.
  Interventions: Device: AcQMap Imaging and Mapping System

INTERVENTIONS:
Device: AcQMap Imaging and Mapping System — 3D Cardiac Imaging and Mapping during ablation procedures
  Other Names: AcQMap

SUMMARY:
A prospective, single-arm, multi-center, multi-national, non-randomized, post-market study designed to provide clinical data regarding the use of the AcQMap High Resolution Imaging and Mapping System during an atrial fibrillation retreatment ablation procedure. (CLP-AF-004 [EU])

A prospective, single-arm, multi-center, non-randomized, pre-market study designed to provide clinical data regarding the use of the AcQMap High Resolution Imaging and Mapping System during an atrial fibrillation retreatment ablation procedure. (CLP-AF-005 [Canada])

DETAILED DESCRIPTION:
A prospective, single-arm, multi-center, multi-national, non-randomized, post-market study designed to provide clinical data regarding the use of the AcQMap High Resolution Imaging and Mapping System during an atrial fibrillation retreatment ablation procedure. The patient population includes men and women, eighteen (18) years of age or older. The treatment plan must include evaluation and ablation (as indicated) of pulmonary vein reconnections plus AcQMap guided non-PV substrate ablation. Subject assessments will occur at screening, procedure, hospital discharge, 3-, 6-, and 12-months. (CLP-AF-004 [EU])

A prospective, single-arm, multi-center, multi-national, non-randomized, pre-market study designed to provide clinical data regarding the use of the AcQMap High Resolution Imaging and Mapping System during an atrial fibrillation retreatment ablation procedure. The patient population includes men and women, eighteen (18) years of age or older. The treatment plan must include evaluation and ablation (as indicated) of pulmonary vein reconnections plus AcQMap guided non-PV substrate ablation. Subject assessments will occur at screening, procedure, hospital discharge, 3-, 6-, and 12-months. (CLP-AF-005 [Canada])

ELIGIBILITY:
Inclusion Criteria:

* Male or female eighteen (18) years of age or older
* Currently scheduled for a repeat endocardial ablation of AF where the index atrial fibrillation ablation procedure was completed ≤ twenty-four (24) months prior to enrollment and the subject has demonstrated at least one episode of post-ablation non-self-terminating AF

Exclusion Criteria:

* No more than two (2) previous left-atrial ablations
* Structural heart disease or implanted cardiac devices
* History of blood clotting or bleeding disease
* Pregnant or lactating (current or anticipated during study follow up)
* Evidence of left atrial thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Grace, MD, Principal Investigator — Papworth Hospital NHS
Locations (14):
- UZ Brussel Centrum voor Hart-en Vaatziekten, Belsele, Jette, Belgium
- Southlake Regional Health Center, Newmarket, Ontario, Canada
- Na Homolce Hospital, Prague, Czechia
- Germany (3):
  - Klinikum Coburg, Coburg
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Netherlands (2):
  - St. Antonius Hospital, Nieuwegein
  - Erasmus MC, Rotterdam
- United Kingdom (6):
  - Papworth Hospital NHS, Cambridge
  - Royal Brompton Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospital Northern, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AcQMap Imaging and Mapping
Started | 128
Treated Subjects | 106 (106 subjects underwent an ablation procedure)
Completed | 103
Not Completed | 25

BASELINE CHARACTERISTICS:
Population: Number of subjects treated
Arm/Group | AcQMap Imaging and Mapping
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 104
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmation of Electrical Isolation of All Pulmonary Veins and Elimination/Modification of All Non-PV Targets
Description: At the procedure conclusion, confirmation of electrical isolation of all pulmonary veins and elimination/modification of all non-PV targets as identified by the AcQMap System
Time Frame: 12 hours
Population: Individual vein isolation was not documented in the protocol. Subjects leaving the lab in sinus rhythm was the surrogate for vein isolation.
Measure: Count of Participants; unit: Participants
Arm/Group | AcQMap Imaging and Mapping
Number analyzed (Participants) | 106
Participants | 99

2. Secondary Outcome: Number of Subjects Who Are Atrial Fibrillation Free at 6 Months Post Procedure
Description: Recording of all subjects who are atrial fibrillation free from events lasting > 30 seconds at 6-months as measured by a 48-hour continuous ECG
Time Frame: 6 months
Population: Subjects who completed a continuous ECG recording at 6-months
Measure: Count of Participants; unit: Participants
Groups:
- AcQMap Arm: Single arm study no randomized control
Arm/Group | AcQMap Arm
Number analyzed (Participants) | 100
Participants | 85

3. Secondary Outcome: Procedure Performance: Total Procedure Time Defined as First Venous Access to Last Cardiac Catheter Out
Description: Documentation of procedure data including total time
Time Frame: 4 hours
Population: Total procedure time defined as first venous access to last cardiac catheter out
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Subjects Completing the AcQMap Procedure: Subjects completing the AcQMap Procedure
Arm/Group | Subjects Completing the AcQMap Procedure
Number analyzed (Participants) | 106
hours | 3.3 (0.8)

4. Secondary Outcome: Procedure Performance: Total Fluoroscopy Time
Description: Documentation of procedure data including fluoroscopy time
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Subjects Completing the AcQMap Procedure
Number analyzed (Participants) | 106
minutes | 25.6 (12.5)

5. Secondary Outcome: Procedure Performance: Ablation Times for PVI
Description: Documentation of procedure data including ablation times for PVI
Time Frame: 2 hours
Population: Total RF ablation time for pulmonary vein isolation
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Subject Who Completed the AcQMap Procedure Receiving Pulmonary Vein Ablations: Subject who completed the AcQMap procedure receiving pulmonary vein ablations
Arm/Group | Subject Who Completed the AcQMap Procedure Receiving Pulmonary Vein Ablations
Number analyzed (Participants) | 76
minutes | 8.5 (6.8)

6. Secondary Outcome: Procedure Performance: Ablation Times for Non-PV Targets
Description: Documentation of procedure data including ablation times for non-PV targets
Time Frame: 2 hours
Population: Total RF ablation time for non-PV triggers
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Subjects Completing the AcQMap Procedure and Receiving Ablations for Non-PV Triggers: Subjects completing the AcQMap procedure and receiving ablations for non-PV triggers
Arm/Group | Subjects Completing the AcQMap Procedure and Receiving Ablations for Non-PV Triggers
Number analyzed (Participants) | 103
minutes | 26.2 (19.3)

7. Secondary Outcome: Number of Subjects Who Are Atrial Fibrillation Free at 12 Months Post Procedure
Description: Recording of all subjects who are atrial fibrillation free from events lasting > 30 seconds at 12-months as measured by a 48-hour continuous ECG
Time Frame: 12 months
Population: Subjects who completed a continuous ECG recording at 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | AcQMap Arm
Number analyzed (Participants) | 103
Participants | 78

ADVERSE EVENTS:
Time Frame: 24-hours post procedure
Arm/Group | AcQMap Imaging and Mapping
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 10/128
Other Adverse Events (participants affected / at risk) | 11/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcQMap Imaging and Mapping (N=128)
Tamponade (Cardiac disorders) | 1 (1)
Urine infection (Renal and urinary disorders) | 1 (1) — Urine infection with urinary retention
Gallstone (Hepatobiliary disorders) | 1 (1) — Gallstone cholecystitis
Arteriovenous fistula (Vascular disorders) | 1 (1)
Atrial groin bleeding (Injury, poisoning and procedural complications) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
ST-Elevation V1-V3 (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1) — Fever after pvi within 48 hours with prolongation
Aneurysm (Vascular disorders) | 1 (1) — Aneurysm spurium right groin
Recurrence of atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AcQMap Imaging and Mapping (N=128)
groin hematoma (Vascular disorders) | 2 (2)
Right groin bleed (Vascular disorders) | 2 (2)
Haematurie (Renal and urinary disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Bi-lateral and right
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Skin Burn (Skin and subcutaneous tissue disorders) | 1 (1)
Suspicion neurological event post procedure (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction of individual site publication until the multi-center data is published

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03368781/Prot_SAP_000.pdf